CLINICAL TRIAL: NCT07088120
Title: PRecision-Controlled Ventilation to Enhance Cardiac Arrest Intervention and Survival IN CPR: A Multi-Center Randomized Controlled Trial
Brief Title: PRECISION-CPR: PRecision-Controlled Ventilation in CPR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Jie Li, Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPR-RCT 001
Record Dates: First submitted 2025-07-10; First posted 2025-07-28 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Arrest (CA)
Keywords: ventilation; tidal volume; cardiac pulmonary resuscitation; real-time feedback; Return of spontaneous circulation
MeSH Terms: conditions — Heart Arrest; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio to either precision-controlled ventilation with real-time feedback or standard ventilation without feedback during CPR. Both groups will be treated concurrently, and outcomes will be compared between groups using a parallel design across multiple centers.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Precision-Controlled Ventilation with Real-Time Feedback (Experimental): Patients will receive manual ventilation during CPR using real-time feedback devices (EOlife) to guide tidal volume (6-8 mL/kg predicted body weight) and ventilation rate (10 breaths per minute) delivery, ensuring adherence to guideline-recommended ventilation parameters.
  Interventions: Device: Precision-Controlled Ventilation with Real-Time Feedback
- Standard of Care Ventilation During CPR (Active Comparator): Patients will receive manual ventilation during CPR per standard practice without real-time feedback, using clinician judgment for tidal volume (visible chest rise) and ventilation rate, consistent with American Heart Association guidelines.
  Interventions: Other: Standard Manual Ventilation During CPR

INTERVENTIONS:
Device: Precision-Controlled Ventilation with Real-Time Feedback — Manual ventilation during CPR using a real-time feedback device (EOlife, Archeon Medical) to guide the delivery of tidal volumes (6-8 mL/kg predicted body weight) and ventilation rate (10 breaths per minute). The device measures and displays ventilation parameters in real time, helping providers achieve guideline-recommended targets during resuscitation.
  Arms: Precision-Controlled Ventilation with Real-Time Feedback
Other: Standard Manual Ventilation During CPR — Manual ventilation during CPR without real-time feedback, using clinician judgment to guide tidal volume (visible chest rise) and ventilation rate, consistent with American Heart Association guidelines.
  Arms: Standard of Care Ventilation During CPR

SUMMARY:
Cardiac arrest is a life-threatening emergency that requires immediate treatment with cardiopulmonary resuscitation (CPR). While chest compressions circulate blood, manual ventilation provides oxygen to the patient. Current CPR guidelines recommend specific ventilation rates and tidal volumes, but studies show that clinicians often deliver too much or too little ventilation due to a lack of monitoring tools, potentially reducing the effectiveness of CPR and impacting survival.

The PRECISION-CPR study is a multi-center, randomized controlled trial designed to evaluate whether using real-time feedback devices to precisely control ventilation during CPR can improve patient outcomes. Adult patients experiencing in-hospital cardiac arrest will be randomized to receive either standard manual ventilation guided by clinician experience or precision-controlled ventilation tailored to the patient's predicted body weight using real-time monitoring devices.

The primary outcome of the study will be return of spontaneous circulation (ROSC). Secondary outcomes will include survival to hospital discharge, neurological recovery, and other clinical measures. By addressing the limitations of current ventilation practices, this study aims to generate evidence to guide future resuscitation guidelines and improve survival rates after cardiac arrest.

DETAILED DESCRIPTION:
The PRECISION-CPR trial is a prospective, multi-center, randomized controlled trial evaluating the effect of precision-controlled ventilation on outcomes during cardiopulmonary resuscitation (CPR) in adult in-hospital cardiac arrest. The study aims to determine whether the use of real-time feedback devices to guide tidal volume (6-8 mL/kg predicted body weight) and respiratory rate (10 breaths per minute) improves return of spontaneous circulation (ROSC) and other clinical outcomes.

Participants are randomized 1:1 to either:

Intervention Group: Manual ventilation guided by real-time feedback device providing continuous tidal volume and respiratory rate feedback during CPR.

Control Group: Manual ventilation performed per standard care without feedback, with the same devices used in blinded mode to record but not display ventilation data.

Ventilation parameters are recorded breath-by-breath. Hemodynamic and clinical variables (e.g., heart rate, end-tidal CO₂) are obtained from the electronic medical record and time-synchronized with ventilation data. Data are collected in REDCap and monitored by a central coordinating center. A Data Safety Monitoring Board oversees safety, protocol adherence, and interim analyses.

The study uses a parallel assignment model and includes stratified randomization by center. Detailed eligibility criteria and outcome measures are recorded in their respective ClinicalTrials.gov sections. The trial is powered to detect differences in ROSC and includes prespecified secondary outcomes and subgroup analyses. The protocol includes quality assurance procedures, interim analyses, and real-time feedback training for clinical teams to ensure intervention fidelity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older) with in-hospital cardiac arrest receiving manual ventilation via bag-mask or artificial airway

Exclusion Criteria:

* Inability to estimate predicted body weight (e.g., extreme body habitus or lack of height data).
* Patients receiving Extracorporeal Membrane Oxygenation (ECMO).
* Known pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Return of Spontaneous Circulation (ROSC) | During resuscitation (up to 60 minutes after cardiac arrest onset)
  Documented presence of a palpable pulse and measurable blood pressure during resuscitation after initiation of CPR.

SECONDARY OUTCOMES:
Survival to Hospital Discharge | Through hospital discharge (up to 28 days after enrollment)
  Survival of the patient to hospital discharge following the index cardiac arrest event during which CPR and the study intervention were delivered.
Neurological Status at Hospital Discharge | At time of hospital discharge (up to 28 days after CPR event)
  Neurological function assessed using the Cerebral Performance Category (CPC) score at the time of hospital discharge, categorized as favorable (CPC 1-2) or unfavorable (CPC 3-5).
Time to Return of Spontaneous Circulation (ROSC) | From initiation of CPR to termination of resuscitation efforts (up to 60 minutes after CPR initiation)
  Time interval from initiation of CPR to achievement of documented ROSC, defined as the presence of a palpable pulse and measurable blood pressure.
Duration of Mechanical Ventilation | From intubation until extubation or hospital discharge, up to 60 days.
  Total number of days the patient receives invasive mechanical ventilation during the index hospitalization following cardiac arrest.
Length of ICU Stay | From ICU admission until ICU discharge, up to 60 days.
  Total length of stay in the intensive care unit during the index hospitalization following cardiac arrest.
New Occurrence of Pneumothorax During CPR | During resuscitation (up to 60 minutes after cardiac arrest onset)
  Incidence of newly diagnosed pneumothorax occurring during CPR and resuscitation efforts, confirmed by clinical assessment and imaging if available.

CONTACTS AND LOCATIONS:
Locations (2):
- Rush University Medical Center, Chicago, Illinois, United States
- Hospital Civil Fray Antonio Alcalde, University of Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD) outside the study team due to institutional policies, data privacy regulations, and the sensitive nature of cardiac arrest data. Aggregate de-identified results will be disseminated through peer-reviewed publications and presentations.

REFERENCES:
- [Background] Kim JW, Park SO, Lee KR, Hong DY, Baek KJ. Efficacy of Amflow(R), a Real-Time-Portable Feedback Device for Delivering Appropriate Ventilation in Critically Ill Patients: A Randomised, Controlled, Cross-Over Simulation Study. Emerg Med Int. 2020 Apr 24;2020:5296519. doi: 10.1155/2020/5296519. eCollection 2020. PMID 32377436
- [Background] Lee ED, Jang YD, Kang JH, Seo YS, Yoon YS, Kim YW, Jeong WB, Ji JG. Effect of a Real-Time Audio Ventilation Feedback Device on the Survival Rate and Outcomes of Patients with Out-of-Hospital Cardiac Arrest: A Prospective Randomized Controlled Study. J Clin Med. 2023 Sep 18;12(18):6023. doi: 10.3390/jcm12186023. PMID 37762963
- [Background] Drennan IR, Lee M, Heroux JP, Lee A, Riches J, Peppler J, Poitras A, Cheskes S. The impact of real-time feedback on ventilation quality during out-of-hospital cardiac arrest: A before-and-after study. Resuscitation. 2024 Nov;204:110381. doi: 10.1016/j.resuscitation.2024.110381. Epub 2024 Sep 18. PMID 39299509
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Alonso A, Beaton AZ, Bittencourt MS, Boehme AK, Buxton AE, Carson AP, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Ferguson JF, Generoso G, Ho JE, Kalani R, Khan SS, Kissela BM, Knutson KL, Levine DA, Lewis TT, Liu J, Loop MS, Ma J, Mussolino ME, Navaneethan SD, Perak AM, Poudel R, Rezk-Hanna M, Roth GA, Schroeder EB, Shah SH, Thacker EL, VanWagner LB, Virani SS, Voecks JH, Wang NY, Yaffe K, Martin SS. Heart Disease and Stroke Statistics-2022 Update: A Report From the American Heart Association. Circulation. 2022 Feb 22;145(8):e153-e639. doi: 10.1161/CIR.0000000000001052. Epub 2022 Jan 26. PMID 35078371
- [Background] Algahtani AI, Scott JB, Li J. Ventilation and Oxygenation During and After Adult Cardiopulmonary Resuscitation: Changing Paradigms. Respir Care. 2024 Nov 18;69(12):1573-1586. doi: 10.4187/respcare.12427. PMID 39288964
- [Background] Scott JB, Schneider JM, Schneider K, Li J. An evaluation of manual tidal volume and respiratory rate delivery during simulated resuscitation. Am J Emerg Med. 2021 Jul;45:446-450. doi: 10.1016/j.ajem.2020.09.091. Epub 2020 Oct 9. PMID 33077312
- [Background] Panchal AR, Bartos JA, Cabanas JG, Donnino MW, Drennan IR, Hirsch KG, Kudenchuk PJ, Kurz MC, Lavonas EJ, Morley PT, O'Neil BJ, Peberdy MA, Rittenberger JC, Rodriguez AJ, Sawyer KN, Berg KM; Adult Basic and Advanced Life Support Writing Group. Part 3: Adult Basic and Advanced Life Support: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S366-S468. doi: 10.1161/CIR.0000000000000916. Epub 2020 Oct 21. No abstract available. PMID 33081529
- [Background] Becker LB, Aufderheide TP, Graham R. Strategies to Improve Survival From Cardiac Arrest: A Report From the Institute of Medicine. JAMA. 2015 Jul 21;314(3):223-4. doi: 10.1001/jama.2015.8454. No abstract available. PMID 26132709
- [Background] Moskowitz A, Grossestreuer AV, Berg KM, Patel PV, Ganley S, Casasola Medrano M, Cocchi MN, Donnino MW; Center for Resuscitation Science. The association between tidal volume and neurological outcome following in-hospital cardiac arrest. Resuscitation. 2018 Mar;124:106-111. doi: 10.1016/j.resuscitation.2017.12.031. Epub 2017 Dec 29. PMID 29292026